CLINICAL TRIAL: NCT01020773
Title: Extubation With or Without Spontaneous Breathing Trial
Acronym: SBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: scientific research office of beijing shijitan hospital, beijing shijitan hospital
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: Beijing Shijitan Hospital
Record Dates: First submitted 2009-03-21; First posted 2009-11-26 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-10

CONDITIONS: Respiratory Failure
Keywords: extubation,Respiration, Artificial
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBT group (Active Comparator): In the SBT group, the patients underwent a 1 hr SBT with inspiratory PS of 7 cmH2O with other settings remaining constant (FiO2, PEEP, trigger sensitivity). The patients who tolerated the SBT underwent immediate extubation.
  Interventions: Behavioral: spontaneous breathing trial
- no-SBT group (No Intervention): In no-SBT group, as soon as a patient met readiness criteria, he or she underwent extubation without SBT process.
  Interventions: Behavioral: spontaneous breathing trial

INTERVENTIONS:
Behavioral: spontaneous breathing trial

SUMMARY:
Spontaneous breathing trial (SBT) has long been thought to be a essential process before extubation. In this study,the investigator hypothesized that SBT could be not essential during weaning from ventilator and investigated whether weaning could be better done without a spontaneous breathing trial in non-COPD（COPD, Chronic Obstructive Pulmonary Disease） critically ill patients. This study has revealed, for the first time, that compared with use of SBT in discontinuing ventilator process, patients underwent successful extubation without SBT. For this subset of patients the findings suggest that SBT may be excluded preceding extubation in a general intensive care population.

DETAILED DESCRIPTION:
In this 1000-bed primary teaching hospital, the study was conducted in the 8-bed adult general ICU over the course of 13 months. All patients enrolled in this study were mechanically ventilated for more than 48 hrs via endotracheal tubes during the study period. The investigation was approved by the hospital ethics committee, and informed written consent was obtained from the next of kin of every patient. Patients were ventilated in pressure support (PS) during the entire weaning period. The levels of inspiratory PS and positive end-expiratory pressure （PEEP) were progressively reduced depending on the patient's clinical assessment and blood gas values. Patients enrolled in this study had to meet all of the following readiness criteria: show significant improvement or resolution of the underlying cause of acute respiratory failure; be fully awake; require bronchial toilet less than twice in the 4 hours proceeding the assessment; stable hemodynamics without further need of vasoactive agents; arterial oxygen tension (PaO2)/fraction of inspired oxygen (FiO2) ratio >200 at a PEEP of 4.0 cm H2O with a maximal FiO2 of 0.40; core temperature <38.0℃; systolic blood pressure >90 mmHg; respiratory rate to tidal volume ratio (RVR) <105 breaths/min/L. The RVR was calculated after 1 min of spontaneous breathing.The maximal inspiratory PS of 12 cm H2O and no mandatory machine breaths supplied from the ventilator.

Study protocol The investigators investigated the weaning process with and without SBT. All patients were continuously assessed according to the readiness criteria and were screened for enrollment once a day. As soon as the patient was ready for weaning, he or she was randomly assigned to SBT or no-SBT study groups. Randomization was carried out in a blinded fashion using opaque and sealed envelopes. All patients in the study breathed through the ventilator circuit with flow-triggering (2L/min) and pressure support ventilation mode. In the SBT group, the patients underwent a 1 hr SBT with inspiratory PS of 7 cmH2O with other settings remaining constant (FiO2, PEEP, trigger sensitivity). For patients showing poor tolerance to the SBT, full ventilation support was immediately recommenced. This was defined by the following failure criteria: a decrease in oxygen saturation to <90%; respiratory rate >35/min for more than 5 min, in the presence of diaphoresis or thoraco-abdominal paradox; sustained increase in heart rate (>140/min), or significant change in systolic blood pressure (>180 or <90 mmHg). The patients who tolerated the SBT underwent immediate extubation and received (breathed in) supplemental oxygen via a facemask. In no-SBT group, as soon as a patient met readiness criteria, he or she underwent extubation without SBT process and received supplemental oxygen via a facemask. Following extubation, noninvasive ventilatory support was introduced in the following circumstances: hypoxemia (SaO2<90% for >15mins) under receiving supplemental oxygen; presence of respiratory acidosis (arterial PH<7.35 with arterial carbon dioxide tension (PaCO2)>45mmHg; and respiratory rate >25 breaths/min for 1 hr. The mode of ventilation was Bi-level Positive Airway Pressure (BiPAP). When such support was deemed inadequate (hypoxemia, hypercapnea, or respiratory distress), the patient was reintubated and mechanically ventilated.

The SBT and extubation were performed by two doctors who are members of the research team. Decisions regarding reintubation were made by doctors who were blinded for the treatment group. Extubation failure is defined as reintubation within 48 hrs. The reasons for reintubation were prospectively recorded.

Statistical Analysis Results are expressed as mean ± SD. Mean values of selected demographic variables and physiologic parameters of patients who underwent SBT were compared by student's t tests to those who underwent extubation directly. The differences in proportions between the two groups were determined using chi square test (X2-test).

ELIGIBILITY:
Inclusion Criteria:

* Mechanically Ventilated patient

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- SBT Group: In the Spontaneous Breathing Trial(SBT) group, the patients underwent a 1 hr SBT with Inspiratory Support Pressure(PS) of 7 cmH2O with other settings remaining constant (FiO2, PEEP, trigger sensitivity). The patients who tolerated the SBT underwent immediate extubation.
Period: Overall Study
Arm/Group | SBT Group | No-SBT Group
Started | 35 | 32
Completed | 31 | 29
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SBT Group | No-SBT Group | Total
Number analyzed (Participants) | 35 | 32 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1.0
  Between 18 and 65 years | 20 | 18 | 38.0
  >=65 years | 15 | 13 | 28.0
Age Continuous [Mean (Standard Deviation); unit: years] | 58.9 (16.3) | 56.7 (18.0) | 57.9 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25.0
  Male | 22 | 20 | 42.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Extubation, Reintubation and in Hospital Mortality
Time Frame: 13 months
Measure: Number; unit: participants
Arm/Group | SBT Group | No-SBT Group
Number analyzed (Participants) | 31 | 29
participants
  Successful extubation | 28 | 29
  Reintubation | 3 | 3
  In hospital mortality | 3 | 4
Statistical Analysis 1: Comparison: SBT Group vs No-SBT Group; Test type: Superiority or Other; p > 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | SBT Group | No-SBT Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No